CLINICAL TRIAL: NCT01146925
Title: A Phase II, Randomized, Double-Blind, Placebo-Controlled Trial to Assess the Efficacy and Safety of CRMD-001 in Contrast-Induced Acute Oxidative Kidney Injury
Brief Title: Deferiprone for the Prevention of Contrast-Induced Acute Kidney Injury
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CorMedix (Industry)
Responsible Party: Robert Hopkins, DVM, MS/Head Clinical Operations and Project Management, CorMedix
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CRMD-001-2001
Record Dates: First submitted 2010-06-16; First posted 2010-06-22 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2011-06

CONDITIONS: Contrast-Induced Acute Kidney Injury
Keywords: Acute Kidney Injury; Contrast-Induced Nephropathy; Labile Iron; Iron Chelation; Deferiprone
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CRMD-001-Deferiprone (Experimental)
  Interventions: Drug: CRMD-001-Deferiprone
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CRMD-001-Deferiprone — CRMD-001 represents unique formulations of Deferiprone. Subjects will be given one (900 mg) immediate release and two (900 mg) extended release tablets 1-3 hours prior to angiography and then every 12 hours for a total of 8 days
  Arms: CRMD-001-Deferiprone
Drug: Placebo — 3 placebo tablets will be given every 12 hours for a total of 8 days, beginning 1-3 hours prior to angiography
  Arms: Placebo

SUMMARY:
The primary objective of this trial is to assess the impact of CRMD-001 on markers of contrast-induced acute kidney injury (AKI) in high-risk patients with chronic kidney disease (CKD) undergoing coronary angiography and PCI.

DETAILED DESCRIPTION:
This trial will evaluate whether treatment with CRMD-001 (unique formulations of the iron chelator, Deferiprone) will reduce the incidence of AKI in subjects with CKD and additional risk factors. Adult subjects with moderate to severe CKD who are undergoing coronary angiography and PCI will be randomized to either placebo or CRMD-001 and followed for 90 days. Subjects will receive 8 days of randomized therapy starting 1-3 hours prior to angiography. The primary endpoint of the trial will be the difference in mean paired change of a panel of sensitive renal biomarkers between the groups. Differences in renal or cardiovascular clinical events will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or older
2. eGFR of < 60 ml/min/1.73 m2
3. Presence of at least one additional risk factor:

   * Diabetes Mellitus
   * Age ≥ 75 years
   * Left Ventricular Ejection Fraction ≤ 40%

Exclusion Criteria:

1. End-Stage Renal Disease
2. Recent change in serum creatinine
3. Primary PCI for STEMI
4. Currently receiving mechanical ventilation
5. Severe heart failure of cardiogenic shock
6. Requirement for inotropic support (prior 30 days)
7. Sustained hypertension > or = 200/110
8. Subject not expected to live for 90 days
9. Anticipated use of ioxaglate or iohexol
10. Currently receiving fenoldopam, dopamine, theophylline, aminophylline, mannitol, N-acetyl cysteine or Ascorbic acid
11. Absolute neutrophil count < 1500
12. Hemoglobin < 8 gm/dL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2010-06; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Biomarker evidence of Acute Kidney injury | 8 Days
  Mean paired change in a panel of acute kidney injury (AKI) biomarkers (urinary NGAL, LFABP, interleukin-18 (IL-18), kidney injury molecule-1 (KIM-1), urinary alpha GST (proximal tubular injury), Pi GST (distal tubular injury) and cystatin C; serum cystatin C) from baseline (Day 1) to peak in the deferiprone and placebo treatment groups, within 192 hours of contrast exposure

SECONDARY OUTCOMES:
Incidence of Acute Kidney Injury | 48 hours
  Incidence of AKI defined as an absolute increase in serum Cr of ≥ 0.3 mg/dL, and/or a 50% relative increase in serum Cr from baseline (Day 1) to a maximum value obtained within 48 hours of contrast exposure

CONTACTS AND LOCATIONS:
Overall Officials: Peter A. McCullough, MD, MPH, Principal Investigator — St. John Providence Health System, Novi, MI
Locations (8):
- United States (8):
  - The Care Group, St. Vincent's Hospital, Indianapolis, Indiana
  - St. John Hospital and Medical Center, Detroit, Michigan
  - Cardiac and Vascular Research Center of Northern Michigan, Petoskey, Michigan
  - Providence Hospital, Southfield, Michigan
  - Ohio Health Research Institute, Columbus, Ohio
  - Cardiovascular Catheterization Labs at Fairfield, Fairfield, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Oklahoma Cardiovascular Research Group, Oklahoma City, Oklahoma